CLINICAL TRIAL: NCT03382067
Title: Influence of Chocolate With Plant Additives on Episodic Memory in Healthy Subjects Experiencing Test Anxiety
Acronym: MaRS-Basel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Prof. Dominique de Quervain, MD, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MaRS-Basel
Record Dates: First submitted 2017-11-23; First posted 2017-12-22 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Test Anxiety

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Epicatechin/ Melissa (Active Comparator): Single consumption of a 55g bar of dark chocolate containing: 42.8g Acticoa ® chocolate + 7.2g caster sugar + 5g Melissa containing 374 mg (-)-Epicatechin/100g chocolate and 2,69% of rosmarinic acid in Melissa leaves
  Interventions: Dietary Supplement: High Epicatechin/ Melissa
- Low Epicatechin/ Oat bran (Placebo Comparator): Single consumption of a 55g bar of white chocolate containing: 50g Lindor ® chocolate + 5g oat bran containing < 0,0009 mg (-)-Epicatechin/100g
  Interventions: Other: Low Epicatechin/ Oat bran

INTERVENTIONS:
Dietary Supplement: High Epicatechin/ Melissa — Single consumption of a 55g bar of dark chocolate containing: 42.8g Acticoa chocolate + 7.2g caster sugar + 5g Melissa
  Arms: High Epicatechin/ Melissa
Other: Low Epicatechin/ Oat bran — Single consumption of a 55g bar of white chocolate containing: 50g Lindor chocolate + 5g oat bran
  Arms: Low Epicatechin/ Oat bran

SUMMARY:
Randomized, blind parallel group design. Single intake of 55 g high Epicatechin /Melissa dark chocolate containing 160 mg Epicatechin per 55 g serving or single intake of 55 g low Epicatechin/ oat bran white chocolate containing < 0,00045 mg Epicatechin per 55 g serving.

A Total of 128 participants, 64 in each group, approx. equal number of male and female. There will be replacement of Drop-Outs until data from 128 participants are completed.

The primary endpoints will be performance in a pictorial memory task and a verbal memory task .

The secondary endpoints will be performance in a working memory test, Saliva cortisol, Visual analog scales assessing, anxiety, confidence, interference, solicitude, and excitement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy by history
* normotensive (BP between 90/60 mmHg and 140/90 mmHg)
* BMI between 18 and < 30 kg/m2
* male or female
* aged between 18 and 30 years
* native or fluent German-speaking
* Prüfungsangstfragebogen (PAF) total or subscale interference score T value > 60

Exclusion Criteria:

* Known hypersensitivity or allergy to cocoa, Melissa, oat, vanillin, milk, soja, nuts
* gluten intolerance
* lactose intolerance
* acute or chronic psychiatric disorder including drug or alcohol abuse
* women who are pregnant or breast feeding
* any clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease etc., infections)
* known or suspected non-compliance
* smoking (> 5 cigarettes per day)
* participation in one of our previous studies using the same memory tests in the past 2 years
* participation in a study with investigational drug within the 30 days preceding and during the present study
* long-term medication within last 3 months (oral contraceptives are disregarded)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Pictorial memory task | 25 minutes and 24 h after presentation
  Participants will be presented with 24 neutral, 24 positive and 24 negative photographs in a random order. Scores will be calculated by summing the correctly remembered photographs per valence.
Verbal memory task | 25 minutes and 24 h after presentation
  Six series of five semantically unrelated nouns will be presented.Total score is calculated by summing the number of correctly recalled words

SECONDARY OUTCOMES:
Saliva cortisol level | 1 day after word/picture presentation Start /middle and end of day. Baseline cortisol 1-14 days later.
  Samples are collected at different timepoints during the day in order to measure stress related cortisol activity. Participants have to chew a cotton sponge for 2-3 minutes, which then are contained in a special device
Working memory | 1 day after word/picture presentation
  Participants will have to calculate as many arithmetical means of seven one-digit numbers possible within two minutes by mental calculation.
Visual Analogue Scale VAS test anxiety | 1 day after word/picture presentation
  will be assessed between each task by the participant using a visual analogue scale. Respondents specify their level of agreement to the statement by indicating a position along a continuous line (10 cm).
Visual Analogue Scale VAS confidence | 1 day after word/picture presentation
  will be assessed between each task by the participant using a visual analogue scale. Respondents specify their level of agreement to the statement by indicating a position along a continuous line (10 cm).
Visual Analogue Scale VAS interference | 1 day after word/picture presentation
  will be assessed between each task by the participant using a visual analogue scale. Respondents specify their level of agreement to the statement by indicating a position along a continuous line (10 cm).
Visual Analogue Scale VAS solicitude | 1 day after word/picture presentation
  will be assessed between each task by the participant using a visual analogue scale. Respondents specify their level of agreement to the statement by indicating a position along a continuous line (10 cm).
Visual Analogue Scale VAS excitement | 1 day after word/picture presentation
  will be assessed between each task by the participant using a visual analogue scale. Respondents specify their level of agreement to the statement by indicating a position along a continuous line (10 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique DeQuervain, Prof. MD, Principal Investigator — University Basel Divison of Cognitive Neuroscience
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No